CLINICAL TRIAL: NCT03108391
Title: A Comparison of the Ambu®AuraGain™ and the Laryngeal Mask Airway Supreme™ in Normal Airway Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Juhui Liu, Plastic Surgery Hospital, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PSH-2016-8
Record Dates: First submitted 2017-03-14; First posted 2017-04-11 (Actual); Last update posted 2017-04-12 (Actual); Status verified 2017-04

CONDITIONS: Supraglottic Airway

STUDY DESIGN:
Intervention Model Description: Parellel Assignment
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ambu AuraGain (Experimental): Subjects will receive the Ambu AuraGain size 3 to size 5 based on manufacturer guidelines
  Interventions: Device: Ambu AuraGain
- LMA Supreme (Active Comparator): Subjects will receive the LMA Supreme size 3 to size 5 based on manufacturer guidelines
  Interventions: Device: LMA Supreme

INTERVENTIONS:
Device: Ambu AuraGain
  Arms: Ambu AuraGain
Device: LMA Supreme
  Arms: LMA Supreme

SUMMARY:
The study is designed to compare the performance of the Ambu AuraGain Laryngeal Mask Airway and LMA Supreme in normal airway patients.

DETAILED DESCRIPTION:
Ambu AuraGain Laryngeal Mask Airway is a newly designed supraglottic device. We design this study to test its clinical performance in normal airway patients, in comparison with LMA Supreme.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists Ⅰ-Ⅲ classification
* Patients evaluated as eligible for a LMA
* Body Mass Index ≤35kg/m2

Exclusion Criteria:

* Patients with known or predicted difficult airway
* Active respiratory infection
* Risk of aspiration
* Head and neck surgery
* Emergent surgery

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-10-31 (Estimated); Study Completion 2017-10-31 (Estimated)

PRIMARY OUTCOMES:
Oropharyngeal leak pressure | Up to 1 minute after the time of confirmed device placement
  The airway pressure at which an airway leak is observed after successful placement of the device

SECONDARY OUTCOMES:
Insertion time | Up to 1 minute on each insertion attempt
  Time needed to insert the device
Ease of insertion | Up to 1 minute on each insertion attempt
  Number of attempts to place the device
Fiberoptic Grade of Laryngeal View | Up to 1 minute after placement of device
  Fiberoptic Grade of Laryngeal View through each device will be graded using a previously grading system
Postoperative Complications | 2 hours after removal of the device
  Patient will be evaluated for sore throat, dysphonia, stridor, dysphagia, blood stain on device

CONTACTS AND LOCATIONS:
Overall Officials: Liu Juhui, MD, Principal Investigator — Plastic Surgery Hospital, ChineseAMS
Locations (1):
- ChineseAMS, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided